CLINICAL TRIAL: NCT06229522
Title: Patients Derived Organoids as a Promising Tool to Tailor Ovarian Cancer Therapies (PANDORA)
Acronym: PANDORA
Status: Recruiting | Type: Observational
Sponsor: Centro di Riferimento Oncologico - Aviano (Other)
Responsible Party: Sponsor
Other Study IDs: CRO-2022-45
Record Dates: First submitted 2023-12-12; First posted 2024-01-29 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The association of clinical, pathogenesis and mutational profile of patients affected by ovarian cancer have improved the armamentarium of therapies available for medical doctors. One of most remarkable advancements is represented by the introduction of PARP inhibitors in the front-line setting of advanced ovarian carcinoma. It is necessary to continue with this effort and introduce novel approaches to improve the survival rate as well as predictive biomarkers to approved therapies. Given the absence of predictive biomarkers to standard therapy, patients derived organoid could be a promising platform to test clinically available drugs and/or promising new molecules to explore the tumor sensibility in an ex-vivo model. The aim of this study is to correlate treatment sensibility measured in tumor derived organoids to clinical sensibility seen in real world patients.

DETAILED DESCRIPTION:
The association of clinical, pathogenesis and mutational profile of patients affected by ovarian cancer have improved the armamentarium of therapies available for medical doctors. One of most remarkable advancements is represented by the introduction of PARP inhibitors in the front-line setting of advanced ovarian carcinoma. It is necessary to continue with this effort and introduce novel approaches to improve the survival rate as well as predictive biomarkers to approved therapies. Given the absence of predictive biomarkers to standard therapy, patients derived organoid could be a promising platform to test clinically available drugs and/or promising new molecules to explore the tumor sensibility in an ex-vivo model. The aim of this study is to correlate treatment sensibility measured in tumor derived organoids to clinical sensibility seen in real world patients.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form;
2. Female sex;
3. Age ≥18 years;
4. Diagnosis of ovarian cancer;
5. Availability of tumor sample or ascites that is planned to be stored in the Institutional Biobank for research purpose

Exclusion Criteria:

1. Patients for which the tumor/ascites biobanking process could compromise the diagnostic assessments;
2. Pregnancy or breast-feeding
3. History of concomitant or previous malignancy in the last 5 years

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include all consecutive women with a diagnosis of ovarian cancer who fit all inclusion/exclusion criteria between the date in which the study is approved and December 2027. Follow-up information will be collected up to 10 years since enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-11-16 (Actual); Primary Completion 2037-12-31 (Estimated); Study Completion 2037-12-31 (Estimated)

PRIMARY OUTCOMES:
To assess if the drugs' sensibility tested in the 3D organoids derived from biopsies could predict the clinical response (PFS) to therapy regimen for each individual ovarian cancer patient. | up to 36 months
  Patients will be divided into two groups based on IC50 level. Difference in PFS probability between patients with high or low IC50 level will be assessed. Progression-free survival (PFS) will be defined as time from enrolment to progression or death whichever comes first
To assess if the drugs' sensibility tested in the 3D organoids derived from ascites fluids could predict the clinical response (PFS) to therapy regimen for each individual ovarian cancer patient. | up to 36 months
  Patients will be divided into two groups based on IC50 level. Difference in PFS probability between patients with high or low IC50 level will be assessed. Progression-free survival (PFS) will be defined as time from enrolment to progression or death whichever comes first
To assess if the drugs' sensibility tested in the 3D organoids derived from biopsies could predict the clinical response (PFI) to therapy regimen for each individual ovarian cancer patient. | up to 36 months
  Patients will be divided into two groups based on IC50 level. Difference in platinum-free interval for platinum salts (PFI) probability between patients with high or low IC50 level will be assessed. PFI will be defined as time from the date of last dose of first line chemotherapy to the date of first recurrence.
To assess if the drugs' sensibility tested in the 3D organoids derived from ascites fluid could predict the clinical response (PFI) to therapy regimen for each individual ovarian cancer patient. | up to 36 months
  Patients will be divided into two groups based on IC50 level. Difference in platinum-free interval for platinum salts (PFI) probability between patients with high or low IC50 level will be assessed. PFI will be defined as time from the date of last dose of first line chemotherapy to the date of first recurrence.

CONTACTS AND LOCATIONS:
Overall Officials: Vincenzo Canzonieri, MD, Principal Investigator — Centro di Riferimento Oncologico di Aviano (CRO) - IRCCS
Locations (1):
- Centro di Riferimento Oncologico (CRO) di Aviano - IRCCS, Aviano, Pordenone, Italy